CLINICAL TRIAL: NCT04691791
Title: Italian Registry of Cardiovascular Magnetic Resonance on Congenital Anomalies of the Coronary Arteries (ITACA-Registry)
Acronym: ITACA
Status: Completed | Type: Observational
Sponsor: ITAB - Institute for Advanced Biomedical Technologies (Other)
Collaborators: Italian Society of Cardiology (Other)
Responsible Party: Principal Investigator, Francesco Bianco, Medical Doctor, ITAB - Institute for Advanced Biomedical Technologies
Other Study IDs: SIC_001
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Congenital Coronary Artery Abnormality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Italian registry of coronary artery abnormalities diagnosed utilizing cardiac magnetic resonance imaging.

DETAILED DESCRIPTION:
Congenital coronary anomalies (ACC) are relatively rare heart disease, in which a congenital defect of origin, course, and term, of one or more epicardial cardiac coronary arteries, is recognized. The global prevalence is estimated at around 0.6-0.7% in the general population, where the most frequent ACCs consist of the anomalous origin of the right coronary artery from the left breast (ARCA), with a prevalence of 0.23%; while the anomalous origin from the Sn coronary artery from the right breast (ALCA) would seem to have a prevalence of 0.03%.

ACCs have often been associated with an increased risk of Sudden Cardiac Death (SCD), especially in athletes. In fact, within this population, ACCs are counted as the second most frequent cause of SCD after hypertrophic cardiomyopathy.

In the general population, the risk of sudden death from ALCA is estimated at around 6.3% at 20 years, while for ARCA it is estimated at around 0.2% at 20 years. The estimated incidence in athletes instead recognizes a range that varies between 0.5 and 13 deaths per 100,000.

Although ACC are therefore recognized as a frequent cause of sudden cardiac death, a recent English study, conducted on a population of 11,168 young footballers, showed a significantly lower incidence than expected: only two coronary anomalies, an ALCA and an ARCA, respectively; the prevalence was therefore 0.002%, at least 10 times lower than expected.

The most common manifestations of ACC are chest pain, palpitations, dizziness and syncope, although more than 50% of patients with ACC are asymptomatic. In the past, these anomalies could only be described at autopsy, while thanks to the enormous developments that the different cardiac imaging modalities have undergone in recent years, ACCs can now also be detected non-invasively. The initial diagnosis is echocardiography, but a confirmation method is necessary (CT, MRI, or coronary angiography), moreover most of the time the finding can be completely incidental and found in the course of examinations conducted for another reason.

This Registry will enroll patients from different sites in Italy (who decided to join the registry within the Italian Society of Cardiology) objectives aiming at establishing the clinical and imaging correlates in patients with congenital anomalies of coronary origin, found or confirmed by cardiac magnetic resonance imaging. As secondary endpoint will be observed subpopulations of patients: 1) in competitive athletes; 2) patients with ventricular ectopic beats (Lown class ≥2).

ELIGIBILITY:
Inclusion Criteria:

* Patients with anomalous origin of the coronaries diagnosed with cardiac magnetic resonance imaging

Exclusion Criteria:

* Patients with known ischemic heart disease
* Patients with coronary atherosclerotic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing cardiac magnetic resonance imaging who have expressed informed consent to data processing, who have a set of images from which the anomalous origin of the coronaries can be diagnosed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Clinical correlates with imaging findings at the cardiac magnetic resonance imaging. | Up to 3 years from the time of the enrollment
  Chest pain, palpitations, sincope and arrhythmias

SECONDARY OUTCOMES:
prevalence of congenital anomalies of coronary origin in specific patient subpopulations: 1) in competitive athletes; 2) patients with ventricular ectopic beats | Up to 3 years from the time of the enrollment
  Prevalence of coronary arteries abnormalities in competitive athletes and patients with ventricular ectopic beats (Lown class ≥ 2).

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bianco, M.D., Principal Investigator — Ospedali Riuniti Ancona
Locations (1):
- Ospedali Riuniti, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheezum MK, Liberthson RR, Shah NR, Villines TC, O'Gara PT, Landzberg MJ, Blankstein R. Anomalous Aortic Origin of a Coronary Artery From the Inappropriate Sinus of Valsalva. J Am Coll Cardiol. 2017 Mar 28;69(12):1592-1608. doi: 10.1016/j.jacc.2017.01.031. PMID 28335843
- [Result] Brothers JA, Frommelt MA, Jaquiss RDB, Myerburg RJ, Fraser CD Jr, Tweddell JS. Expert consensus guidelines: Anomalous aortic origin of a coronary artery. J Thorac Cardiovasc Surg. 2017 Jun;153(6):1440-1457. doi: 10.1016/j.jtcvs.2016.06.066. Epub 2017 Feb 4. No abstract available. PMID 28274557
- [Result] Eckart RE, Scoville SL, Campbell CL, Shry EA, Stajduhar KC, Potter RN, Pearse LA, Virmani R. Sudden death in young adults: a 25-year review of autopsies in military recruits. Ann Intern Med. 2004 Dec 7;141(11):829-34. doi: 10.7326/0003-4819-141-11-200412070-00005. PMID 15583223
- [Result] Basso C, Maron BJ, Corrado D, Thiene G. Clinical profile of congenital coronary artery anomalies with origin from the wrong aortic sinus leading to sudden death in young competitive athletes. J Am Coll Cardiol. 2000 May;35(6):1493-501. doi: 10.1016/s0735-1097(00)00566-0. PMID 10807452
- [Result] Maron BJ, Doerer JJ, Haas TS, Tierney DM, Mueller FO. Sudden deaths in young competitive athletes: analysis of 1866 deaths in the United States, 1980-2006. Circulation. 2009 Mar 3;119(8):1085-92. doi: 10.1161/CIRCULATIONAHA.108.804617. Epub 2009 Feb 16. PMID 19221222
- [Result] Malhotra A, Dhutia H, Finocchiaro G, Gati S, Beasley I, Clift P, Cowie C, Kenny A, Mayet J, Oxborough D, Patel K, Pieles G, Rakhit D, Ramsdale D, Shapiro L, Somauroo J, Stuart G, Varnava A, Walsh J, Yousef Z, Tome M, Papadakis M, Sharma S. Outcomes of Cardiac Screening in Adolescent Soccer Players. N Engl J Med. 2018 Aug 9;379(6):524-534. doi: 10.1056/NEJMoa1714719. PMID 30089062
- [Result] Villa AD, Sammut E, Nair A, Rajani R, Bonamini R, Chiribiri A. Coronary artery anomalies overview: The normal and the abnormal. World J Radiol. 2016 Jun 28;8(6):537-55. doi: 10.4329/wjr.v8.i6.537. PMID 27358682